CLINICAL TRIAL: NCT01522521
Title: Phase 3 Study of AK156 in Primary Osteoporosis Patients
Brief Title: Study of AK156 in Primary Osteoporosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK156 III-1
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
Keywords: AK156
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1. (Experimental)
  Interventions: Drug: AK156
- 2. (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK156 — zoledronic acid (i.v.)/year + daily calcium and vitamin D for 2 years
  Arms: 1.
Drug: Placebo — placebo (i.v.)/year + daily calcium and vitamin D for 2 years
  Arms: 2.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of AK156 in Japanese patients with primary osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary osteoporosis
* Patients who have vertebral fractures at the time of screening

Exclusion Criteria:

* Patients diagnosed with secondary osteoporosis
* Patients with a current uncontrolled medical disorder or other condition which makes the patient unsuitable for the study

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
New vertebral fractures | 2 Years
  Reduction in the incidence rate of new fragility vertebral fractures

SECONDARY OUTCOMES:
Vertebral fractures (worsening and new) | 2 Years
  The incidence rate of fragility vertebral fractures (worsening and new)
Clinical fractures | 2 Years
  The incidence rate of Clinical fractures
Bone mineral density | 2 Years
  The percent change from baseline in bone mineral density of lumbar spine and hip
Bone metabolic marker | 2 Years
  The percent change from baseline in bone metabolic marker

CONTACTS AND LOCATIONS:
Overall Officials: Asahi Kasei Pharma Corporation, Study Director — Clinical Development Center
Locations (20):
- Japan (20):
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Kure, Hiroshima
  - Sapporo, Hokkaido
  - Inami-cho, Hyōgo
  - Morioka, Iwate
  - Kagoshima, Kagoshima-ken
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Sendai, Miyagi
  - Miyazaki, Miyazaki
  - Matsumoto, Nagano
  - Bungo-ōno, Oita Prefecture
  - Tosu, Saga-ken
  - Tokorozawa, Saitama
  - Kikukawa, Shizuoka
  - Oyama, Tochigi
  - Setagaya City, Tokyo
  - Shinagawa, Tokyo
  - Tonami, Toyama

REFERENCES:
- [Derived] Shiraki M, Kuroda T, Takeuchi Y, Sugimoto T, Tanaka S, Suzuki H, Hiraishi K, Nakamura T. Acute Phase Reactions After Intravenous Infusion of Zoledronic Acid in Japanese Patients with Osteoporosis: Sub-analyses of the Phase III ZONE Study. Calcif Tissue Int. 2021 Dec;109(6):666-674. doi: 10.1007/s00223-021-00884-7. Epub 2021 Jul 10. PMID 34247263
- [Derived] Taguchi A, Shiraki M, Tanaka S, Ohshige H, Nakamura T. Improved periodontal disease and prevention of tooth loss in osteoporosis patients receiving once-yearly zoledronic acid: a randomized clinical trial. Menopause. 2019 Nov;26(11):1277-1283. doi: 10.1097/GME.0000000000001393. PMID 31688575
- [Derived] Nakamura T, Fukunaga M, Nakano T, Kishimoto H, Ito M, Hagino H, Sone T, Taguchi A, Tanaka S, Ohashi M, Ota Y, Shiraki M. Efficacy and safety of once-yearly zoledronic acid in Japanese patients with primary osteoporosis: two-year results from a randomized placebo-controlled double-blind study (ZOledroNate treatment in Efficacy to osteoporosis; ZONE study). Osteoporos Int. 2017 Jan;28(1):389-398. doi: 10.1007/s00198-016-3736-y. Epub 2016 Sep 8. PMID 27631091